CLINICAL TRIAL: NCT03547726
Title: Physical Therapy After Reverse Total Shoulder Arthroplasty: A Randomized Clinical Trial
Brief Title: Physical Therapy After Reverse Total Shoulder Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Amit Momaya, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F11223344
Record Dates: First submitted 2018-04-29; First posted 2018-06-06 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: There will be two groups of patients randomized either to receive formal physical therapy in clinic or a self-led at home rehabilitation regimen.
Who Masked: Care Provider, Investigator
Masking Description: The physician will not know if the patient is receiving at home physical therapy or seeing a physical therapist in clinic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Therapy (Active Comparator): This group of patients will receive a predetermined physical therapy regimen with guidance from a physical therapist.
  Interventions: Other: Physical Therapy
- Self-Rehab (Experimental): This group of patients will be provided with a list of actions not to perform during the stages of their rehab (to avoid injury), and allowed to rehab their shoulder at their own pace.
  Interventions: Other: Self-Rehab

INTERVENTIONS:
Other: Physical Therapy — These patients will receive a formal physical therapy protocol by seeing a physical therapist in clinic.
  Arms: Physical Therapy
Other: Self-Rehab — These patients will be provided with a list of actions NOT to perform and allowed to self rehabilitate. They will not see a physical therapist.
  Arms: Self-Rehab

SUMMARY:
A common operation for various shoulder conditions is a total shoulder arthroplasty (TSA). In cases with severe rotator cuff tears or other conditions, a variant of the procedure called a reverse total shoulder arthroplasty may be performed. It is unclear whether or not patients require formal physical therapy (as opposed to no physical therapy with recommended avoided movements) after reverse TSA. Orthopaedic surgeons have varying opinions on the postoperative rehabilitation protocol for reverse TSA, with some surgeons not prescribing any physical therapy. The purpose of this study is to randomize patients into two groups: one that sees a physical therapist after their reverse TSA, and one that is provided with actions not to perform and are allowed to self-rehabilitate.

DETAILED DESCRIPTION:
A common operation for various shoulder conditions is a total shoulder arthroplasty (TSA). In cases with severe rotator cuff tears or other conditions, a variant of the procedure called a reverse total shoulder arthroplasty may be performed. It is unclear whether or not patients require formal physical therapy (as opposed to no physical therapy with recommended avoided movements) after reverse TSA. Orthopaedic surgeons have varying opinions on the postoperative rehabilitation protocol for reverse TSA, with some surgeons not prescribing any physical therapy. The purpose of this study is to randomize patients into two groups: one that sees a physical therapist after their reverse TSA, and one that is provided with actions not to perform and are allowed to self-rehabilitate.

There is very limited orthopaedic literature focusing on the postoperative rehabilitation after reverse TSA. The majority of research is in the physical therapy literature focusing on the actual rehabilitation protocol. However, there has never been a large, randomized clinical trial that asks the question of whether or not physical therapy after reverse TSA is even necessary, or if patients will have comparable outcomes if they perform their own at home rehabilitation. There are surgeons nationwide that are on either end of the spectrum. Some encourage patients to see a therapist for a prolonged period of time with a set regimen of exercises, while others do not encourage any formal physical therapy and instead give patients a list of movements not to perform and allow them to recover at their own pace. We hypothesize that there will be comparable clinical outcomes between patients randomized to receive physical therapy versus an at home, self-led rehabilitation protocol. There are no deleterious effects of either treatment wing.

Patients who agree to undergo reverse TSA after a preoperative appointment with their attending surgeon will be invited to participate in the study. They will complete the below mentioned survey instruments. They will receive their procedure and appropriate postoperative treatment. Patients will then be randomized to either the physical therapy or self-rehab group. Both groups will receive the standard postoperative physical therapy protocol. The only difference between the groups will be if a physical therapist sees the patients in their clinic, or if the patients self-rehabilitate with a list of limitations throughout their recovery course. The physical therapy protocol provided to the physical therapists and patients is attached.

Clinical outcomes will be measured using the attached survey instruments: Simple Shoulder Test (SST), American Shoulder and Elbow Surgeons Shoulder Score (ASES-SS), and the Single Assessment Numeric Evaluation score (SANE). These are commonly used, validated survey instruments in the setting of orthopaedic shoulder research.

The physical exam component of the study will include range of motion testing (measuring the degrees of movement using a goniometer) and strength testing (measured using the dynamometer) in both shoulders.

These survey instruments and measurements will be performed at 3, 6, and 12 month postoperative follow up.

ELIGIBILITY:
Inclusion Criteria:

* • Patients who agree to receive a reverse total shoulder arthroplasty by one of our participating surgeons

Exclusion Criteria:

* • Revision shoulder replacement surgery

  * Mentally incompetent to provide informed consent
  * Non-english speaking
  * Minors (<18)
  * Pregnant women
  * Prison population
  * Acute Shoulder Fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
Forward Flexion Range of Motion 1 | 3 months followup
  Active range of motion in the shoulder joint in forward flexion (measured in degrees)

SECONDARY OUTCOMES:
Strength 1 | 3 months followup
  Strength measured using a dynamometer
Simple Shoulder Test Patient Reported Outcome 1 | 3 months followup
  12 question questionnaire, scores are 0-12, 12 is best score (normal)
Strength 2 | 6 month followup
  Strength measured using a dynamometer
Strength 3 | 12 months followup
  Strength measured using a dynamometer
Internal Rotation Range of Motion 1 | 3 months followup
  Active range of motion in the shoulder joint in internal rotation (measured in degrees)
External Rotation Range of Motion 1 | 3 months followup
  Active range of motion in the shoulder joint in external rotation (measured in degrees)
Internal Rotation Range of Motion 2 | 6 month followup
  Active range of motion in the shoulder joint in internal rotation (measured in degrees)
External Rotation Range of Motion 2 | 6 month followup
  Active range of motion in the shoulder joint in external rotation (measured in degrees)
Forward Flexion Range of Motion 2 | 6 months followup
  Active range of motion in the shoulder joint in forward flexion (measured in degrees)
Forward Flexion Range of Motion 3 | 12 months followup
  Active range of motion in the shoulder joint in forward flexion (measured in degrees)
Internal Rotation Range of Motion 2 | 12 months followup
  Active range of motion in the shoulder joint in internal rotation (measured in degrees)
External Rotation Range of Motion 2 | 12 months followup
  Active range of motion in the shoulder joint in external rotation (measured in degrees)
American Shoulder and Elbow Surgeons Shoulder Score 1 | 3 month followup
  17 question questionnaire, normalized to a 0-100 scale, 100 is normal
Simple Shoulder Test Patient Reported Outcome 2 | 6 month followup
  12 question questionnaire, scores are 0-12, 12 is best score (normal)
Simple Shoulder Test Patient Reported Outcome 3 | 12 month followup
  12 question questionnaire, scores are 0-12, 12 is best score (normal)
Single Assessment Numeric Evaluation (SANE) Score 1 | 3 month followup
  1 question questionnaire asking to rate overall shoulder function, scores can be 0-100, 100 is optimal score/normal shoulder
American Shoulder and Elbow Surgeons Shoulder Score 2 | 6 month followup
  17 question questionnaire, normalized to a 0-100 scale, 100 is normal
American Shoulder and Elbow Surgeons Shoulder Score 3 | 12 month followup
  17 question questionnaire, normalized to a 0-100 scale, 100 is normal
Single Assessment Numeric Evaluation (SANE) Score 2 | 6 month followup
  1 question questionnaire asking to rate overall shoulder function, scores can be 0-100, 100 is optimal score/normal shoulder
Single Assessment Numeric Evaluation (SANE) Score 3 | 12 month followup
  1 question questionnaire asking to rate overall shoulder function, scores can be 0-100, 100 is optimal score/normal shoulder

CONTACTS AND LOCATIONS:
Overall Officials: Amit M Momaya, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Hospital Highlands, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided